CLINICAL TRIAL: NCT05781633
Title: A Single-arm, Open-label， Phase Ⅱ Clinical Trial of Eutideron, Etoposide Combined With Bevacizumab for Breast Cancer Patients With Brain Metastases
Brief Title: The Efficacy and Safety of Eutideron, Etoposide, and Bevacizumab in Patients With Brain Metastases From Breast Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTD-1-BM-II
Record Dates: First submitted 2023-02-19; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Mammary Neoplasms, Human
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- eutidrone+ etoposide+ bevacizumab (Experimental): Eligible patients received a regimen of eutidrone(30mg/m2/d,iv,d1-5,21d/cycle), etoposide(30mg/m2/d,iv,d1-3,21d/cycle), and bevacizumab (10mg/kg,d1,21d/cycle).At least 4 to 6 cycles were administered, and if patients had a response or stable disease, bevacizumab was used as maintenance therapy until disease progression or intolerable toxicity.
  Interventions: Drug: eutidrone etoposide bevacizumab

INTERVENTIONS:
Drug: eutidrone etoposide bevacizumab — Eligible patients received a regimen of eutidrone(30mg/m2/d,iv,d1-5,21d/cycle), etoposide(30mg/m2/d,iv,d1-3,21d/cycle), and bevacizumab (10mg/kg,d1,21d/cycle).At least 4 to 6 cycles were administered, and if patients had a response or stable disease, bevacizumab was used as maintenance therapy until disease progression or intolerable toxicity.MRI of the brain with contrast enhancement was performed at baseline and every 6 weeks after enrollment; thereafter, patients with stable disease or a response could be assessed at a reduced frequency to every 9 weeks; central nervous system and noncentral nervous system lesions were assessed according to RANO-BM criteria and RECIST v1.1 criteria until disease progression, respectively.

SUMMARY:
This study was a single-arm, open-label, phase II study of breast cancer patients with brain metastases. Eligible patients received a regimen of eutidrone(30mg/m2/d,iv,d1-5,21d/cycle), etoposide(30mg/m2/d,iv,d1-3,21d/cycle), and bevacizumab (10mg/kg,d1,21d/cycle).At least 4 to 6 cycles were administered, and if patients had a response or stable disease, bevacizumab was used as maintenance therapy until disease progression or intolerable toxicity.

DETAILED DESCRIPTION:
The natural survival time of breast cancer patients with brain metastases is short and the prognosis is poor. Although the treatment is progressing, but it is still limited. The current domestic guidelines still recommend local therapy as a priority treatment strategy. At the same time, about 80% of patients with brain metastasis will progress to extracranial metastasis, so superior systemic treatment is particularly important, but very lacking.Therefore, new systematic therapeutic drugs are urgently needed .Eutiderone is a new generation of epirubicin anti-tumor drug with good efficacy and safety. In pre-clinical studies, it has been shown that the drug concentration in most tissues is higher than that in plasma, and the concentration of eutiderone in brain tissue is higher, indicating that the drug is easy to cross the blood-brain barrier.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Female,>18.
* Histologically or cytologically confirmed recurrent metastatic breast cancer.
* ECOG:0-2.
* There was at least one measurable lesion in the central nervous system.
* Based on screening brain magnetic resonance imaging (MRI), patients with CNS must meet one of the following conditions：
* Untreated brain metastases from breast cancer do not require immediate local treatment.
* Previously treated breast cancer brain metastases that have progressed after previous central nervous system local treatment as assessed by the investigator and that do not have clinical features requiring immediate local treatment.
* Previous anti-HER2 therapy and TKI therapy were required for HER2+ patients.
* Patients who had not received chemotherapy, radiotherapy, surgery, targeted therapy or immunotherapy within 4 weeks before enrollment.
* All toxicity in patients associated with previous antitumor therapy must be restored to ≤ grade 1 (CTCAE v5.0). However, patients with any grade of alopecia were allowed.
* Routine blood tests were normal within 1 week before enrollment (according to the normal range at the participating laboratory):White blood cell count (WBC) ≥ 3.0 × 109/L; Neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 100 × 109/L; Hemoglobin ≥ 9.0 g/dL; patients could receive blood transfusions or erythropoietin to meet this criterion.
* Liver and kidney function were basically normal within 1 week before enrollment (based on the normal values of the participating laboratory):Total bilirubin (TBIL) ≤ 2.5× upper limit of normal value (ULN); Alanine aminotransferase (SGPT/ALT) ≤2.5×ULN (≤5×ULN in patients with liver metastases); Aspartate aminotransferase (SGOT/AST) ≤2.5×ULN (≤5×ULN in patients with liver metastases); Creatinine clearance (Ccr) ≥60 ml/min
* Male or female patients of childbearing potential had to consent to use an effective method of contraception, such as dual barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc., during the study period and up to 90 days after the last study medication was taken. Female patients of reproductive age had to have a negative blood or urine pregnancy test before enrollment.
* Life expectancy ≥ 12 weeks.

Exclusion Criteria:

* Other malignant tumors (including primary brain or leptomeningeal related tumors) within the past 5 years, except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
* Previous anti-tumor therapy, including chemotherapy, radical radiotherapy, hormone therapy, biological therapy, immunotherapy or anti-tumor traditional Chinese medicine therapy within 4 weeks before initiation of study treatment.
* Patients had previously used eutidrone injection, etoposide, or bevacizumab.
* Patients had undergone major organ surgery (excluding needle biopsies) or major trauma within 4 weeks before the first dose of the study drug, or required elective surgery during the trial.
* Patients with ≥grade 3 neurosystem-related severe adverse reactions after previous use of anti-microtubules.
* Patients with any untreated > 2.0cm brain injury, unless discussed with the investigator and approved for registration.
* Systemic corticosteroids were continued to control symptoms of brain metastases at a total daily dose of >2mg dexamethasone (or equivalent). However, patients with chronic stable doses ≤2mg daily of dexamethasone (or equivalent) may be discussed and approved by the investigator.
* Any brain lesion deemed to require immediate local treatment, including (but not limited ) increased lesion size at anatomical sites or possible treatment-related edema, may pose a risk to the patient (e.g.brain stem lesions). Patients received local treatment were still eligible for study based on lesions identified by screening contrast brain MRI according to the criteria described in the CNS inclusion criteria.
* More than 2 seizures within 4 weeks before enrollment.
* Poor control of hypertension; Or a previous history of hypertensive crisis or hypertensive encephalopathy.
* Patients had a history of hemoptysis within 6 months before enrollment. Or evidence of bleeding tendency or significant coagulopathy within the past 1 month.
* Currently receiving full-dose warfarin or equivalent, or aspirin (325mg/ day) within 10 days
* The need for major surgery, open biopsy, or major trauma was anticipated within 28 days or during the course of the study.
* Patients with a history of abdominal fistula or gastrointestinal perforation within the previous 6 months; The presence of an unhealed wound, active ulcer, or untreated fracture; Pregnant or lactating women.
* Patients with a history of psychotropic drug abuse and inability to abstain or with mental disorders.
* Other nonmalignant systemic diseases (cardiovascular, renal, liver, etc.) that were treated by any treatment regimen or prevented follow-up were excluded.
* Known or suspected allergies to any of the study drugs or excipients.
* No brain MRI for any reason.
* Any other condition considered by the investigator to be unsuitable for participation in the trial.
* Other situations in which corticosteroid use is prohibited.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 43 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
CNS Objective response rate (CNS-ORR) | 12 months
  The proportion of patients with complete response (CR) and partial response (PR) evaluated as the best response observed from enrollment to progression of all CNS target lesions assessed according to RANO-BM criteria among the total number of patients who could be evaluated.

SECONDARY OUTCOMES:
CNS Clinical benefit rate(CNS-CBR) | 3 months
  Percentage of patients who achieved complete response (CR), partial response (PR), or stable disease (SD) in all CNS target lesions assessed by RANO-BM criteria within 12 weeks.
CNS Progression-free survival (CNS-PFS) | 36 months
  Time from enrollment to the first radiographic documented disease progression (PD) of all CNS target lesions (RANO-BM criteria) or death from any cause without progression was recorded.
Objective response rate (ORR) | 12 months
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
Progression-free survival（PFS） | 36 months
  Time from enrollment to the first radiographically confirmed disease progression (PD) (RECIST 1.1 criteria) or death from any cause without documented progression
Overall survival (OS) | 36 months
  Time from the enrollment to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yehui Shi, MD,Phd, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Yehui Shi, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No